CLINICAL TRIAL: NCT02254174
Title: A Randomised, Open-label Four-way Crossover Study to Evaluate Relative Bioavailability of Tiotropium and Salmeterol After Inhalation of a Fixed Combined Single Dose (7.5 μg Tiotropium, 25 μg Salmeterol, Inhalation Powder, Hard Capsule, HandiHaler®2), a Free Combined Single Dose of 18 μg Tiotropium [Spiriva® HandiHaler®] and 50 μg Salmeterol [Serevent® Diskus®], a Single Dose of 50μg Salmeterol (Serevent® Diskus®) and a Single Dose of 18 μg Tiotropium (Spiriva® HandiHaler®) in Healthy Male Volunteers
Brief Title: Relative Bioavailability of Tiotropium and Salmeterol After Inhalation of a Fixed Combined Dose Compared to Monocomponents in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1184.11
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Tiotropium Bromide; Salmeterol Xinafoate

ARMS (4):
- Tiotropium/Salmeterol (Experimental)
  Interventions: Drug: Tiotropium/Salmeterol
- Serevent® Diskus® (Active Comparator)
  Interventions: Drug: Serevent® Diskus®
- Spiriva® (Active Comparator)
  Interventions: Drug: Spiriva®
- Spiriva® and Serevent® Diskus® (Active Comparator)
  Interventions: Drug: Serevent® Diskus®; Drug: Spiriva®

INTERVENTIONS:
Drug: Tiotropium/Salmeterol — Fixed dose combination of tiotropium 7.5 μg and salmeterol 25 μg inhalation powder, PE capsule via HandiHaler®
  Arms: Tiotropium/Salmeterol
Drug: Serevent® Diskus®
  Arms: Serevent® Diskus®; Spiriva® and Serevent® Diskus®
Drug: Spiriva®
  Arms: Spiriva®; Spiriva® and Serevent® Diskus®

SUMMARY:
Assessment of the relative bioavailability of a fixed dose combination of tiotropium and salmeterol compared to a free dose combination of the marketed products of tiotropium and salmeterol (Spiriva® and Serevent® Diskus®).

Assessment of the relative bioavailability of a fixed dose combination of tiotropium and salmeterol compared to tiotropium and salmeterol administered as individual mono substances from the marketed products.

Assessment of safety and tolerability of the fixed combination of tiotropium and salmeterol in a PE (Polyethylene) capsule administered via the HandiHaler® 2

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male based upon a complete medical history, including the physical examination, regarding vital signs (blood pressure (BP), pulse rate (PR)), 12-lead ECG (electrocardiogram) measurement, and clinical laboratory tests. There is no finding deviating from normal and of clinical relevance.

   There is no evidence of a clinically relevant concomitant disease
2. Age ≥21 and ≤50 years
3. BMI ≥18.5 and <30 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR, and ECG measurements) deviating from normal and of clinical relevance
2. Evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of relevant allergy/hypersensitivity (including allergy to the drug or its excipients) as judged clinically relevant by the investigator
8. Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to randomisation
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to enrolment in the study or during the study
10. Participation in another trial with an investigational drug within 2 months prior to randomisation
11. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
12. Inability to refrain from smoking on trial days as judged by the investigator
13. Alcohol abuse (more than 40 g alcohol a day)
14. Drug abuse
15. Blood donation (more than 100 mL blood within 4 weeks prior to randomisation or during the trial)
16. Excessive physical activities within 1 week prior to randomisation or during the trial
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of the study centre

    The following exclusion criteria are specific for this study due to the known class side effect profile of ß2-mimetics:
19. Asthma or history of pulmonary hyperreactivity
20. Hyperthyrosis
21. Allergic rhinitis in need of treatment
22. Clinically relevant cardiac arrhythmia
23. Paroxysmal tachycardia (>100 beats per minute)

    The following exclusion criteria are specific for this study due to the known class side effect profile of tiotropium:
24. Hypersensitivity to tiotropium and/or related drugs of this class

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-03; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of salmeterol in blood plasma over the time interval from 0 extrapolated to infinity); | Up to 8 hours after drug administration
Cmax (maximum measured concentration of salmeterol in blood plasma) | Up to 8 hours after drug administration
Ae0-8 (urinary excretion of tiotropium over an 8 hour interval) | Up to 8 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve in plasma over the time interval from 0 to the time of the last quantifiable data point) | Up to 8 hours after drug administration
AUC0-∞ (area under the concentration-time curve of tiotropium in blood plasma over the time interval from 0 extrapolated to infinity) | Up to 8 hours after drug administration
Cmax (maximum measured concentration of tiotropium in blood plasma) | Up to 8 hours after drug administration
AUCt1-t2 (area under the concentration time curve in plasma over the time interval t1 to t2) | up to 8 hours after inhalation
tmax (time from dosing to the maximum concentration of in plasma) | Up to 8 hours after drug administration
λz (terminal rate constant in plasma) | Up to 8 hours after drug administration
t½ (terminal half-life of in plasma) | Up to 8 hours after drug administration
MRTih (mean residence time in the body after inhalational administration) | Up to 8 hours after drug administration
CL/F (apparent clearance of in the plasma after extravascular administration) | Up to 8 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | Up to 8 hours after drug administration
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2 | up to 8 hours after inhalation
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 8 hours after inhalation
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 8 hours after inhalation
Number of participants with abnormal findings in physical examination | up to 90 days after first drug administration
Number of participants with clinically significant changes in vital signs | up to 90 days after first drug administration
Number of participants with abnormal findings in 12-lead ECG | up to 90 days after first drug administration
Number of participants with abnormal changes in clinical laboratory parameters | up to 90 days after first drug administration
Number of participants with adverse events | up to 90 days after first drug administration
Tolerability assessed by investigator on a 4-point scale | up to 90 days after first drug administration